CLINICAL TRIAL: NCT04383158
Title: Characterisation of Wound Healing in the Dental Extraction Socket With and Without Plasma Rich in Growth Factors (PRGF). A Pilot Study
Brief Title: Alveolar Socket Healing With and Without PRGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 279109
Record Dates: First submitted 2020-05-01; First posted 2020-05-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Bone Resorption; Wound Heal
Keywords: alveolar ridge preservation; autologous platelet concentrates; 3-D; randomised controlled study; plasma rich in growth factors; PRGF; Dental Implants

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, single-centre, prospective, parallel-group qualitative pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRGF extraction sockets (Test) (Active Comparator): Immediately after dental extraction, the socket will be filled with Plasma Rich in Growth Factors (ENDORET® POST-EXTRACTION ALVEOLUS DENTAL KIT (KMU16))
  Interventions: Other: PRGF ENDORET® obtained from ENDORET® POST-EXTRACTION ALVEOLUS DENTAL KIT (KMU16)
- Unassisted extraction sockets (Control) (No Intervention): Dental extraction sockets to be left to heal spontaneously unassisted.

INTERVENTIONS:
Other: PRGF ENDORET® obtained from ENDORET® POST-EXTRACTION ALVEOLUS DENTAL KIT (KMU16) — ENDORET® POST-EXTRACTION ALVEOLUS DENTAL KIT (KMU16) is a system for obtaining plasma rich in growth factors (PRGF), which can be applied in the regeneration of bone and other connective tissues in oral surgery. PRGF is a completely autologous blood platelet concentrate that stimulates tissue regeneration due to enrichment with autologous growth factors, acting as a biological system.
  Arms: PRGF extraction sockets (Test)

SUMMARY:
A single-centre randomised controlled pilot study involving 12-24 healthy adult patients for investigating dental extraction socket healing with and without plasma rich in growth factors (PRGF) taking place during early days of healing (days 1, 3, 7, 15, 30) and relating the healing to clinical and histological outcomes after 90 days of healing. Healing will be investigated by means of various non-invasive imaging technologies (e.g. laser scanners, thermal cameras, laser cameras) in addition to conventional technologies (e.g. bone core biopsy, 3D xray images). At 90 days of healing, dental implants will be placed in the healed sockets and implants will be restored and followed up until 12 months after connecting the prosthesis to the implant (e.g. implant crown). Dental implant outcomes (e.g. survival, success) will also be evaluated.

DETAILED DESCRIPTION:
Randomised, controlled, single-centre, prospective, parallel-group qualitative pilot study. Objectives: the study aims to characterise wound healing events in the dental extraction socket with and without plasma rich in growth factors (PRGF) taking place during early days of healing after a dental extraction and their relation to clinical and histological outcomes after 90 days of healing. The early healing events of the post-extraction socket will be characterized in terms of volumetric changes in relation to intra-oral thermographic changes, blood flowgraphy, molecular (proteomic) changes, as well as extra-oral integrated geometric thermographic changes in tandem with clinical measures of soft tissue healing, post-operative pain assessment. The early healing events will be analysed in relation to volumetric, clinical and histomorphometric changes of new bone formation after 90 days of healing during dental implant treatment. Dental Implant outcomes will be evaluated up to 12 months after loading.

Duration: Overall, we anticipate that the study will last approximately 28 months. We estimate a 3-month study set-up period, followed by a recruitment period of 6 months. Each participant will attend 14 visits over approximately 18-19 months. The first 9 visits involve a dental extraction and follow-up until 90 days after extraction to obtain a bone core biopsy and dental implant placement. Visits 10 to 14 will be for restoring the dental implant and evaluating dental implant treatment outcomes.

ELIGIBILITY:
Inclusion Criteria

All of the following criteria must be fulfilled for inclusion:

* Patient must have willingness to read and sign a copy of the Informed Consent Form Males and females, ≥25 years old.
* Patient in need of a single permanent tooth extraction with clinical and/or radiographic evidence of unrestorable maxillary premolars, canines, or incisors with at least one adjacent tooth present, and with periodontal attachment preserved at least for 2/3rd of the root nor associated with acute periapical pathology.
* Post-extraction alveolar bone defect with ≤50 % buccal bone loss. This will be confirmed at Visit 2 after extraction. In case of >50% buccal bone loss, the participant will be withdrawn.
* Patient in good general health as documented by self-assessment.
* Full mouth bleeding and plaque scores (FMBS <10% and FMPS <20%) recorded within the previous 8 weeks.

Exclusion criteria

* Uncontrolled or untreated periodontal disease.
* History of local (head and neck) radiation therapy.
* Presence of oral lesions in the area of the extraction (such as ulceration, malignancy).
* Severe bruxing or clenching habits.
* Acute endodontic lesion in the test tooth or in the neighbouring areas to the extraction procedure (sites with presence of an asymptomatic chronic lesion are eligible).
* Medical history that includes uncontrolled diabetes or hepatic or renal disease, or other serious medical conditions that can impact on bone metabolism (e.g. rheumatoid arthritis, osteoporosis) or transmittable diseases (e.g. AIDS).
* History of alcohol or drug abuse.
* Smokers.
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* Malocclusion, or collapse of the occlusal vertical dimension leading to dentoalveolar compensation which could interfere with ridge preservation dimensions and measurements.
* Lack of adjacent sound restored or unrestored teeth.
* Any male participants with facial hair (such as moustache, beard or any other variations of facial hair styles) and must keep their face shaven until after the placement of the dental implant (Visit 10).
* Any individuals using Botox or fillers in the face region.

All patients to be enrolled who meet the inclusion / exclusion criteria will be asked if they have participated in any other interventional periodontal studies within the last 3 months. If the patient did participate in such studies, then enrolment will be postponed until after 3 months wash-out period has elapsed.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Intra-oral geometric and thermographic changes of the alveolar ridge | From dental extraction and post-operative days 1, 3, 7, 15, 30 and 90.
  Changes expressed as percentages of intra-oral geometric volumes and temperatures within a defined region of interest (ROI) at 1, 3, 7, 15, 30 and 90 days after dental extraction in unassisted socket healing and PRGF-assisted healing. The ROIs will include the buccal, crestal, and palatal surfaces of the extraction socket defined proximally between two vertical planes parallel to the tooth axis in the middle of the mesial and distal papilla, and defined superiorly by a horizontal plane at the level of the mucogingival line.dental extraction in unassisted socket healing and PRGF-assisted healing.

SECONDARY OUTCOMES:
Extra-oral geometric changes of the whole face at 1, 3, 7, 15, and 30 days after dental extraction | From dental extraction and post-operative days 1, 3, 7, 15, and 30.
  Changes expressed as percentages of extra-oral geometric volumes at selected areas of interest at 1, 3, 7, 15, and 30 days after dental extraction
Extra-oral thermographic changes of the whole face at 1, 3, 7, 15, 30 and 90 days after dental extraction | From dental extraction and post-operative days 1, 3, 7, 15, 30 and 90.
  Changes expressed as percentages of extra-oral thermographic changes at selected areas of interest at 1, 3, 7, 15, 30 and 90 days after dental extraction.
Blood flowgraphy changes of intra-oral soft tissue of the dental extraction socket | From dental extraction and post-operative days 1, 3, 7, 15, 30 and 90.
  Changes expressed as percentage of blood flowgraphy measured with Laser Speckle Contrast Imaging (LSCI) of intra-oral soft tissue of the dental extraction socket
Molecular (proteomic) changes of wound exudate of the dental extraction socket | From dental extraction and post-operative days 1, 3, 7, and 15.
  Descriptive account of molecular (proteomic) changes of wound exudate of the dental extraction socket after extraction based on the Normalised Spectral Abundance Factor (NSAF) proteomic analysis
Clinical changes of the intra-oral soft tissue of the dental extraction socket measured by soft tissue healing index of Landry (Landry, 1985) | From dental extraction and post-operative days 1, 3, 7, and 15.
  Qualitative clinical changes of the intra-oral soft tissue of the dental extraction socket measured by soft tissue healing index of Landry (Landry, 1985)
Post-operative pain assessed with a visual analogue scale (VAS) | From dental extraction and post-operative days 1, 3, 7, and 15.
  Changes in the values of reported visual analogue scale (VAS) of 10 grades (value of 1= no pain, value of 10= maximum pain) to assess post-operative pain
Geometric changes of 3-D radiographic bone (CBCT) and 3-D optically scanned soft tissue at suture removal (7 days) and at 90 days of healing | At suture removal at 7 days after dental extraction and at 90 days of healing.
  Percentage of geometric changes of 3-D radiographic bone (CBCT) and 3-D optically scanned soft tissue at suture removal (7 days) and at 90 days of healing
Histomorphometric new bone formation assessed with histology and X-ray microtomography (XMT), to calculate the percentages of new bone within bone core samples obtained after 3 months of healing at the dental implant placement procedure | At 90 days of healing after dental extraction.
  Percentage of new bone formation assessed with histological analysis and X-ray microtomography (XMT) within bone core samples obtained after 3 months of healing at the dental implant placement procedure
Feasibility of implant placement expressed as percentages (%) of implants placed with satisfactory primary stability | At 90 days of healing after dental extraction.
  Percentage of implants placed with satisfactory primary stability in the optimal prosthetically driven 3-D position
Need for further augmentation expressed as a percentage (%) of implants that required further ridge augmentation procedures during implant placement for the management of residual dehiscence or fenestration defects | At 90 days of healing after dental extraction.
  Percentage of implants that required further ridge augmentation procedures during implant placement for the management of residual dehiscence or fenestration defects
Implant survival and success according to success criteria of Buser et al (Buser et al., 1990) assessed at 12 months after implant loading | At 12 months after implant loading
  Percentage of implant survival and success according to success criteria of Buser et al (Buser et al 1990)
- Molecular (proteomic) changes of the peri-implant crevicular fluid at suture removal after implant placement and at 6 months and 12 months after implant loading | at suture removal after implant placement and at 6 months and 12 months after implant loading.
  - Descriptive account of molecular (proteomic) changes of the peri-implant crevicular fluid at suture removal after implant placement and at 6 months and 12 months after implant loading
Papilla Fill Index, Pink Esthetic Score (PES) and White Esthetic Score (WES) at 6 months and 12 months after implant loading | at 6 months and 12 months after implant loading
  PFI, PES and WES scores
- Intra-oral geometric changes of the peri-implant soft tissue at 6 months and 12 months after implant loading | at 6 months and 12 months after implant loading
  Percentage of geometric changes of the peri-implant soft tissues

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, DDS, MS, PhD, Principal Investigator — Centre for Oral Clinical Research, Institute of Dentistry, Barts & The London School of Medicine & Dentistry, QMUL
Locations (1):
- Centre for Oral Clinical Research, London, United Kingdom